CLINICAL TRIAL: NCT00802152
Title: Using Health Information Technology (HIT) to Improve Ambulatory Chronic Disease Care: Smart Device Substudy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1095618
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Hypertension; Diabetes
Keywords: Diabetes; Hypertension
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Monitoring (Experimental): 100 eligible subjects identified as (HbA1c >= 8% OR SBP > 130 mm Hg)
  Interventions: Other: Home monitoring
- Usual Care (No Intervention): 100 eligible subjects identified as (HbA1c >= 8% OR SBP > 130 mm Hg)

INTERVENTIONS:
Other: Home monitoring — The subject will take their blood pressure or glucose measurements 1-4 times per day, depending on patient condition. They will upload these measurements using the device to a secure website at least every other day. Data will be reviewed at least 2 times per week Monday through Friday by the clinic nursing staff. Data indicating problems, e.g., critical out of range values, will be communicated to the patient's primary care physician after review by the nurse. The physician will then determine what is needed for follow up action based on the patient's condition and data (e.g., telephone call to patient home, scheduling a clinic appointment, etc).
  Other Names: MetrikLink, MediCompass, iMetrikus
  Arms: Home Monitoring

SUMMARY:
In-home health monitoring devices have the potential to increase the speed and ease of modifying treatment for ambulatory patients living with chronic conditions. This study examines the implementation and effectiveness of remote data transmission from in-home devices (blood glucose meter/blood pressure machine) to the clinic on treatment outcomes in patients with diabetes who have out of range blood glucose (BG) or systolic blood pressure (BP) measurements. We test whether the short-term targeted use of in-home monitoring devices facilitates management for providers and improves outcome measures for patients.

DETAILED DESCRIPTION:
To evaluate the effectiveness of short-term targeted use of remote data transmission from in-home devices (blood glucose meter/blood pressure machine) to the clinic on treatment outcomes in patients with diabetes who have out of range blood glucose (BG) or systolic blood pressure (BP) measurements. Increased frequency of data transmission will provide the provider with "real time" data in order to make more timely adjustments in the treatment plan, resulting in improved glycemic control as measured by A1c values and hypertension as measured by systolic blood pressure (SBP).

Subjects will be recruited from Family & Community Medicine (FCM) and General Internal Medicine (GIM) clinics. We will randomly select patients from physicians with a minimum number of 5 eligible patients from the performance measurement list (A1c>=8% or SBP>130) to approach for the study. Patients who agree to enroll will be randomized to experimental and control using a block randomization approach stratified by age increments (18-40; 41-55; 56-70; 71+). Subjects will be randomized using prepared sealed envelopes. A total of 200 subjects (100 intervention subjects and 100 control subjects) will be enrolled over a period of one year. We will attempt to enroll equal numbers of FCM and GIM subjects.

For all subjects, baseline data will be collected from the patient, including demographic data (age, gender, race, and years of formal education), payor status (private pay, insurance, Medicaid), number of co-morbid conditions, baseline blood pressure, and length of time diagnosed with diabetes (DM) and hypertension.

Intervention patients will be instructed to test their BP and BG according to a minimum protocol of at least once daily and upload this clinical data at least every other day for the 3-month study duration, but this frequency could be further tailored by their provider, i.e., more than once daily. At least 2 of these BG readings each week should be fasting levels. Patient training will emphasize that this system is not an emergency response system, i.e., critical values should be treated in the usual manner.

Control group patients (those who do not receive the device) will be asked to test their BP and BG at least once daily (in the same fashion as the intervention group). They will be instructed to bring these readings to their clinic visits, and again at the end of the study. We will collect these readings.

Data from patients are downloaded to the website as they enter data. These data may be printed out for MD review or verbally communicated. APNs in FCM will make changes in patient treatment based on their currently established privileges, e.g., medication adjustments; RNs in GIM or FCM will review data with MDs for changes in treatment plans. All treatment changes will be individualized according to patient need, i.e., no standardized blood glucose management protocol will be employed. Communication of changes in therapy to the patient will be accomplished per usual clinic protocol, e.g., usually by a telephone call to the patient, with documentation of a telephone note in the medical record.

After three months, all subjects will return to the clinic for an A1c and BP measure, and for post study surveys. Data collection will include achievement of clinical goals in blood glucose (A1c measure at end of 3 month intervention [+/- 2 weeks] and BP). If enrolled subjects have an available A1c and BP measure recorded in the record at the end of 6 months, we will collect these data to assess longer term effects of the intervention. Patient records will be reviewed for interventions provided to patient (i.e., documenting the process of medication changes, advice provided).

Interview data will be collected from physicians and nurses re: perceptions of use of the data from the device; patient perceptions of the home-device application, and patient use rates of data upload (intervention), and frequency of BG and BP testing both before and during the intervention period (for both intervention and control patients).

The primary outcome measure will be a comparison of A1c at three months following enrollment (i.e., patient met goal of > 0.5% change in A1c or SBP < 130). The proportion of patients who meet the blood glucose / BP goal three months after enrollment will be computed for both the intervention group and the control group. For each group, the denominator will be the number of patients enrolled in that group (and thus were not meeting the recommended goals at the time of enrollment). The numerator will be those patients who meet the recommended goals as determined during an office visit which occurs three months (+/- 14 calendar days) after enrollment.

Changes in care processes will be categorized and described, and related to the patient entered data (daily blood glucose measures).

Physician and nurse perception data will be analyzed using qualitative approaches. Intervention group patient perceptions and satisfaction with the home-device application will be measured using a short survey and analyzed descriptively.

In the intervention group, patient use rates will be calculated to include the percent of readings submitted as the numerator and total expected as denominator (e.g., submitted 70 readings/90 days = 78% use rate).

RN time per week for data review & follow up will be analyzed descriptively to assess the burden of responding to monitoring data.

Data will be collected on the time for enrollment and patient training in order to estimate costs associated with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* hemoglobin A1c (A1c) ≥8% OR systolic BP> 130 on last measurement
* on oral medication or insulin
* Type 2 diabetes
* Diabetes and hypertension for at least one year
* using/owns a blood glucose meter (that is compatible with study equipment)
* followed by an attending MD
* private land phone line or computer with internet connection
* enrolled at Family & Community Medicine (FCM) Green Meadows , FCM Woodrail or Fairview General Internal Medicine (GIM) clinic and anticipate receiving primary care for next 12 months from MU primary care

Exclusion Criteria:

* newly diagnosed or Type 1 diabetes
* legally blind
* currently reside in a long-term care facility, including assisted living facility, residential care
* severe cognitive impairment (6-item cognitive screen via recruitment telephone call)
* family/household member enrolled in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) or Systolic blood pressure (SBP) | Baseline, 3 months

SECONDARY OUTCOMES:
Changes in care (process), abstracted from patient's medical record | 3 months, 6 months following enrollment
Patient-entered device data | All data over three months

CONTACTS AND LOCATIONS:
Overall Officials: David Mehr, MD, Principal Investigator — University of Missouri, School of Medicine
Locations (1):
- University of Missouri, Dept. of Family and Community Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No